CLINICAL TRIAL: NCT03710408
Title: Adverse Effects of Subcutaneous vs Intravenous Hydration on Older Acutely Admitted Patients: An Assessor-blinded, Non-inferiority RCT
Brief Title: Subcutaneous vs Intravenous Hydration on Older Adults
Acronym: SCIV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University Hospital (Other)
Collaborators: Aalborg University (Other)
Responsible Party: Principal Investigator, Mathias Aalkjær Brix Danielsen, Principal Investigator, Aalborg University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: N-20180014
Record Dates: First submitted 2018-06-13; First posted 2018-10-18 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Dehydration
Keywords: Hypodermoclysis; Older adults; Geriatric patient; Hydration therapy; Adverse effects; Subcutaneous hydration
MeSH Terms: conditions — Dehydration | interventions — Hypodermoclysis

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: To achieve assessor/care provider blinding, all participants will receive a sham needle (opposite of the randomization). This will not pierce the skin but just lay on top of the skin. Both the randomized and the sham needle will be covered by non-woven swabs before placement of the dressing. Both the active and the sham device is connected to an infusion set. The infusion tubes will be tangled at the top, just below the roller ball and drop counter. The entanglement will be covered by opaque dressing. This way it cannot be know which infusions tube is connected to the fluid bag, while it is still possible to control the infusion speed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Subcutaneous hydration (Experimental)
  Interventions: Other: Subcutaneous hydration
- Intravenous hydration (Active Comparator)
  Interventions: Other: Intravenous hydration

INTERVENTIONS:
Other: Intravenous hydration — Participants assigned to the intravenous hydration arm will receive their hydration therapy through an intravenous access. This access will be achieved by inserting a "BD VenflonTM Pro Safety - 22G" in a vein in the dorsal side of the hand or further up the forearm. If the participants is suspected of becoming delirious and at risk of removing the cannula from the hand/forearm, it may be inserted at the dorsal side of the foot. The clinical staff judge this risk and decide site of placement.
  Furthermore, a sham subcutaneous access device "BD Saf-T-Intima™ Integrated Safety Catheter System" will be placed on the abdomen without piercing the skin.
  Other Names: BD VenflonTM Pro Safety - 22G
  Arms: Intravenous hydration
Other: Subcutaneous hydration — Participants assigned to the subcutaneous hydration arm will receive their hydration therapy through a subcutaneous access. This access will be achieved by placing a "BD Saf-T-Intima™ Integrated Safety Catheter System" on the abdomen or, alternatively if the participants is suspected of becoming delirious and at risk of removing the needle, it will be placed on the back at the scapular region.
  Furthermore, a sham IV access device "BD VenflonTM Pro Safety - 22G" will be placed on the dorsal side of the hand without piercing the skin.
  Other Names: BD Saf-T-Intima™ Integrated Safety Catheter System
  Arms: Subcutaneous hydration

SUMMARY:
This study will evaluate the risk of adverse effects of intravenous hydration compared to subcutaneous hydration. Half of the patients will receive hydration by the subcutaneous route the other half by the intravenous route. In the subsequent 24 hours period the patients will be monitored for any sign of adverse effects.

DETAILED DESCRIPTION:
Adequate hydration is essential to humans, and is tightly regulated in the healthy adult by in- and output (i.e. thirst and urine production). This regulation is often hampered in the geriatric patient due to a decreased sensation of thirst and impaired kidney function. The risk of dehydration increases rapidly in the acutely ill geriatric patient with the growing fluid demand of fever and reduced ability to self-hydrate due to fatigue. Dehydration will often aggravate an acute illness creating a vicious circle. External rehydration is essential to stop or even prevent this downward spiral. Adequate hydration can be maintained or achieved by two different routes: oral intake or parenteral infusion. When oral hydration is insufficient, intravenous (IV) fluid infusion is the commonly used route. However, subcutaneous (SC) infusion of fluid, also known as hypodermoclysis, is an alternative route.

Several studies have compared SC hydration to IV hydration with the main outcome being laboratory test of hydration or subjective assessment scores. They all found similar effects on laboratory markers of hydration, which align with the theory of mass conservation. They also found a similar incidence of side effects between IV and SC hydration as secondary outcomes. The main drawback of these studies is methodological shortcomings. The lack of blinding introduces a large risk of bias on subjective outcome such as assessment scores and grading of side effects. Furthermore, the largest of the studies had a third of their patients switch groups diluting the result. A recent Cochrane review on achieving parenteral hydration found that the quality of included trials was low and future trials should prospectively register, have secure allocation concealment, adequate sample sizes and should be reported according to established standard.

This study will examine if subcutaneous (SC) hydration is a safe alternative to intravenous (IV) hydration in the geriatric patient in the Emergency Department, Acute Assessment Unit or Orthopedic Ward of Aalborg University Hospital. This will be achived by preforming an assessor-blinded, non-inferior, randomized controlled trial.

Relevant participants (see Eligibility Criteria) arriving at Aalborg University Hospital will be enrolled after informed consent. Baseline measurements will be obtained, and the participants will be randomized (1:1) to either intravenous or subcutaneous hydration. A sham setup will be use so both an intravenous access and a subcutaneous access will be visible on the patient, but only one of them will be active. For the next 24 hours the participants will regularly be evaluated by a nurse blinded to infusion for the presence of adverse effects.

ELIGIBILITY:
Inclusion Criteria:

1. Medical patients admitted to Acute Assessment Unit (AAU). (All internal medicine patients are admitted here first, except highly specialized patients (e.g. ketoacidosis or severe cardiology conditions).
2. Orthopedic hip fracture patients admitted to the orthopedic ward.
3. Patients admitted to short term care.
4. Prescription of 0.5-2 liters of parenteral fluid over the next 24 hours.

Exclusion Criteria:

1. Red triage tag (severe ill patients)
2. Prescription of IV antibiotics or other treatment administrate intravenous
3. Severe dehydration (fluid requirements over 2 liters over 24 hours)
4. Known strict fluid restriction (cannot receive ½ liters of fluid infusion)
5. Severe general edema
6. Unable to give informed consent

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 51 (Actual)
Dates: Start 2019-01-20 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2020-11-01 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse effects (dichotomous variable, blinded, non-inferior) | The participants will be observed for 24 hours after the start of infusion.
  The incidence of adverse effects of hydration therapy (both serious and minor adverse effects) is the primary outcome measure of this study.
  Serious adverse effects will be defined as any consequence of infusion requiring treatment(e.g. diuretics, analgesic and antibiotics)
  Minor adverse effects will be defined as any of the following:
  * Reddening of the skin at infusion site larger than what is covered by dressing.
  * Painful swelling at infusion site.
  * Prolonged swelling at infusion site (more than two hours after end of infusion).
  * Itching.
  * Phlebitis without needing treatment.
  * Patient complaining of infusion related pain.
  * Failure of infusion.
  * Need of reinserting the infusion needle.
  * Accidental catheter removal by the patient.
  * Need for reducing of flow speed due to complaint from the patient.
  Swelling at infusion site, without discomfort or need for action, will not be evaluated as an adverse effect.

SECONDARY OUTCOMES:
Incidence of serious adverse effects (total number of serious adverse effects (discrete variable, blinded) | The participants will be observed for 24 hours after the start of infusion
  A sensitivity analysis of the primary outcome comparing only the serious adverse effects.
Incidence of adverse effects (dichotomous variable, blinded, superiority calculation) | The participants will be observed for 24 hours after the start of infusion.
  Same description as primary outcome, but this calculation will only be performed if non-inferiority is found.
Incidence of adverse effects (total number of adverse effects (discrete variable, not blinded) | The participants will be observed for 24 hours after the start of infusion.
  Same as description primary outcome but this is a comparison of the number of adverse effects the average patient experience.
Personal graded time spend on insertion of active device (ordered categorical variable, non-blinded). | During procedure.
  Nurses will estimate the time of insertion of the active device into the following categories: 1) less than 3 min., 2) 3-5 min, 3) 5-10 min, 4) 10-20 min. If the primary nurse cannot achieve access it will be noted if 5) another ER nurse or an 6) anesthesiological nurse is needed. Lower is better.
Participants evaluation of pain during inserting the active device (continuous variable, non-blinded). | During procedure.
  Participants will evaluate the pain of having the active access device inserted on a Visual Analog Scale (VAS) 0-100 mm. Lower is better.
Participants evaluation of pain during fluid infusion through the active device (continuous variable, non-blinded) | Participants will evaluate this at the end of observation (24 hours after inclusion)
  Participants will evaluate the pain during infusion (24 hours) on a Visual Analog Scale (VAS) 0-100 mm. Lower is better. This will be done for both the active and sham device.
Presence of delirium (dichotomous variable, blinded) | Duration of observation (24 hours)
  Number of delirious participants at end of observation adjusted for number of delirious participants at inclusion. The presence of delirium will be evaluated using Confusion Assessment Method (CAM).
Death during hospitalization (dichotomous variable, blinded) | From inclusion to end of current admission. Cutoff is one month after inclusion.
  Compare death during hospitalization between groups. Both deaths during the observation period and after the end of observation but still during the same admission.

OTHER OUTCOMES:
Effect of infusion method on hydration status, evaluated by P-albumin (continuous variables) | Changes from inclusion to end of observation (24 hours)
  A comparison of changes in albumin. We will refrain from performing statistical analysis on the effect of hydration. This is both due to the complexity of evaluating dehydration status on geriatric patients, but also to avoid a type 1 error due to multiple comparisons.
Effect of infusion method on hydration status, evaluated by P-creatinine (continuous variables) | Changes from inclusion to end of observation (24 hours)
  A comparison of changes in creatinine. We will refrain from performing statistical analysis on the effect of hydration. This is both due to the complexity of evaluating dehydration status on geriatric patients, but also to avoid a type 1 error due to multiple comparisons.
Effect of infusion method on hydration status, evaluated by eGFR (continuous variables) | Changes from inclusion to end of observation (24 hours)
  A comparison of changes in eGFR. We will refrain from performing statistical analysis on the effect of hydration. This is both due to the complexity of evaluating dehydration status on geriatric patients, but also to avoid a type 1 error due to multiple comparisons.
Effect of infusion method on hydration status, evaluated by P-urea (continuous variables) | Changes from inclusion to end of observation (24 hours)
  A comparison of changes in urea. We will refrain from performing statistical analysis on the effect of hydration. This is both due to the complexity of evaluating dehydration status on geriatric patients, but also to avoid a type 1 error due to multiple comparisons.
Effect of infusion method on hydration status, evaluated by P-osmolality (continuous variables) | Changes from inclusion to end of observation (24 hours)
  A comparison of changes in osmolality. We will refrain from performing statistical analysis on the effect of hydration. This is both due to the complexity of evaluating dehydration status on geriatric patients, but also to avoid a type 1 error due to multiple comparisons.
Effect of infusion method on hydration status, evaluated by hemoglobin (continuous variables) | Changes from inclusion to end of observation (24 hours)
  A comparison of changes in hemoglobin. We will refrain from performing statistical analysis on the effect of hydration. This is both due to the complexity of evaluating dehydration status on geriatric patients, but also to avoid a type 1 error due to multiple comparisons.
Effect of infusion method on hydration status, evaluated by P-sodium (continuous variables) | Changes from inclusion to end of observation (24 hours)
  A comparison of changes in sodium. We will refrain from performing statistical analysis on the effect of hydration. This is both due to the complexity of evaluating dehydration status on geriatric patients, but also to avoid a type 1 error due to multiple comparisons.
Effect of infusion method on hydration status, evaluated by P-potassium (continuous variables) | Changes from inclusion to end of observation (24 hours)
  A comparison of changes in potassium. We will refrain from performing statistical analysis on the effect of hydration. This is both due to the complexity of evaluating dehydration status on geriatric patients, but also to avoid a type 1 error due to multiple comparisons.
Effect of infusion method on hydration status, evaluated by blood pressure (both systolic and diastolic will be measured and compared) (continuous variables). | Changes from inclusion to end of observation (24 hours)
  A comparison of changes in blood pressure. We will refrain from performing statistical analysis on the effect of hydration. This is both due to the complexity of evaluating dehydration status on geriatric patients, but also to avoid a type 1 error due to multiple comparisons.

CONTACTS AND LOCATIONS:
Overall Officials: Mathias B Danielsen, MD, Principal Investigator — Aalborg University Hospital
Locations (1):
- Aalborg University Hospital, Aalborg, Denmark

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification. Data sets will only be share where anonymity of included participants can be insured.
Supporting Information: Study Protocol, Analytic Code
Time Frame: Beginning 6 months and ending 5 years following article publication.
Access Criteria: Data will be shared upon reasonable request.

REFERENCES:
- [Background] O'Keeffe ST, Lavan JN. Subcutaneous fluids in elderly hospital patients with cognitive impairment. Gerontology. 1996;42(1):36-9. doi: 10.1159/000213768. PMID 8641599
- [Background] Challiner YC, Jarrett D, Hayward MJ, al-Jubouri MA, Julious SA. A comparison of intravenous and subcutaneous hydration in elderly acute stroke patients. Postgrad Med J. 1994 Mar;70(821):195-7. doi: 10.1136/pgmj.70.821.195. PMID 8183752
- [Background] Slesak G, Schnurle JW, Kinzel E, Jakob J, Dietz PK. Comparison of subcutaneous and intravenous rehydration in geriatric patients: a randomized trial. J Am Geriatr Soc. 2003 Feb;51(2):155-60. doi: 10.1046/j.1532-5415.2003.51052.x. PMID 12558710
- [Background] Ker K, Tansley G, Beecher D, Perner A, Shakur H, Harris T, Roberts I. Comparison of routes for achieving parenteral access with a focus on the management of patients with Ebola virus disease. Cochrane Database Syst Rev. 2015 Feb 26;2015(2):CD011386. doi: 10.1002/14651858.CD011386.pub2. PMID 25914907
- [Derived] Danielsen MB, Worthington E, Karmisholt JS, Moller JM, Jorgensen MG, Andersen S. Adverse effects of subcutaneous vs intravenous hydration in older adults: An assessor-blinded randomised controlled trial (RCT). Age Ageing. 2022 Jan 6;51(1):afab193. doi: 10.1093/ageing/afab193. PMID 34651171

DOCUMENTS (1):
  • Statistical Analysis Plan (2019-08-19): https://cdn.clinicaltrials.gov/large-docs/08/NCT03710408/SAP_000.pdf